CLINICAL TRIAL: NCT06730841
Title: Dose-Optimized and Spaced Transcranial Direct Current Stimulation for Treatment-Resistant Depression
Acronym: DOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jean-Philippe Miron, Assistant Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 810432
Record Dates: First submitted 2024-08-23; First posted 2024-12-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-12

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- DOS-tDCS: A dose-optimized and spaced form of tDCS (Active Comparator): On each treatment day, participants will receive 5 tDCS sessions, each lasting 20 minutes, with a 20-minute intersession interval. The dose-optimized and spaced tDCS (DOS-tDCS) group will be treated using a stimulation intensity of up to 4 mA.
  Interventions: Device: Dose-Optimized and Spaced Transcranial Direct Current Stimulation
- Spaced tDCS: A spaced form of tDCS only (Active Comparator): On each treatment day, participants will receive 5 tDCS sessions, each lasting 20 minutes, with a 20-minute intersession interval. The spaced tDCS only group will receive stimulation at the standard 2 mA dose.
  Interventions: Device: Spaced Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): On each treatment day, participants will receive 5 sham tDCS sessions, each lasting 20 minutes, with a 20-minute intersession interval.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Dose-Optimized and Spaced Transcranial Direct Current Stimulation — tDCS, a non-invasive neuromodulation technique that applies low-intensity, direct electrical stimulation to the cortex via scalp electrodes, has been extensively researched as a potential treatment for MDD. tDCS enhances neuroplasticity, which is theorized to be responsible for its therapeutic effects and has been presented as a cost-effective solution for MDD. Preclinical evidence supports the potential advantage of spaced stimulation with tDCS to maximally engage neuroplasticity. This group will be treated using a stimulation intensity of up to 4 milliamp (mA).
  Participants will first complete an acute intensive induction phase consisting of daily treatment every weekday over 2 weeks (10 days total) followed by a consolidation phase consisting of weekly treatments (once a week) over 4 additional weeks (6 weeks total).
  Other Names: tDCS; Soterix Medical 1x1 CT
  Arms: DOS-tDCS: A dose-optimized and spaced form of tDCS
Device: Spaced Transcranial Direct Current Stimulation — tDCS, a non-invasive neuromodulation technique that applies low-intensity, direct electrical stimulation to the cortex via scalp electrodes, has been extensively researched as a potential treatment for MDD. tDCS enhances neuroplasticity, which is theorized to be responsible for its therapeutic effects and has been presented as a cost-effective solution for MDD. Preclinical evidence supports the potential advantage of spaced stimulation with tDCS to maximally engage neuroplasticity. This group will be treated using a stimulation intensity of 2 mA.
  Participants will first complete an acute intensive induction phase consisting of daily treatment every weekday over 2 weeks (10 days total) followed by a consolidation phase consisting of weekly treatments (once a week) over 4 additional weeks (6 weeks total).
  Other Names: Soterix Medical 1x1 CT
  Arms: Spaced tDCS: A spaced form of tDCS only
Device: Sham Transcranial Direct Current Stimulation — tDCS, a non-invasive neuromodulation technique that applies low-intensity, direct electrical stimulation to the cortex via scalp electrodes, has been extensively researched as a potential treatment for MDD. tDCS enhances neuroplasticity, which is theorized to be responsible for its therapeutic effects and has been presented as a cost-effective solution for MDD. This group will be treated using sham stimulation.
  Participants will first complete an acute intensive induction phase consisting of daily treatment every weekday over 2 weeks (10 days total) followed by a consolidation phase consisting of weekly treatments (once a week) over 4 additional weeks (6 weeks total).
  Other Names: Soterix Medical 1x1 CT
  Arms: Sham tDCS

SUMMARY:
This study aims to evaluate the feasibility, safety, and tolerability of an innovative approach to treating Major Depressive Disorder (MDD), particularly in cases where patients have not responded well to traditional therapies. Specifically, the objective is to evaluate the antidepressant effects of a Dose-Optimized and Spaced Transcranial Direct Current Stimulation (DOS-tDCS) protocol in participants with treatment-resistant depression (TRD) compared to spaced tDCS only and sham tDCS in a 3-arm randomized controlled trial (RCT). The proposed method involves applying low-intensity electrical currents through the scalp in a manner that is both more intense and more frequently spaced than standard treatments. This approach is hypothesized to lead to a significant reduction in depressive symptoms. Participants in the study will be randomly assigned to one of three groups: the experimental group receiving the DOS-tDCS treatment, a group receiving spaced tDCS only, or a control group receiving a sham (placebo) treatment. Outcomes will be measured over a period of six weeks. The study's goal is to offer a potentially more accessible and effective treatment option for individuals who have not benefited from existing MDD therapies.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. People between the ages of 18 and 85 at the time of screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questionnaires / follow instructions during interventions. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
3. Currently diagnosed with Major Depressive Disorder (MDD) and meets criteria for a Major Depressive Episode, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
4. Medical records confirming a history of at least moderate treatment-resistance as defined an Antidepressant Treatment History Form (ATHF) score for that antidepressant trial of > 2 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF score of 1 or 2 on those 2 separate antidepressants) OR have a combination of one failed trial and one not tolerated trial, per the definitions above.
5. MADRS score of ≥20 at screening (Visit 1).
6. Existing relationship with mental health provider and access to ongoing psychiatric care before and after completion of the study.
7. Must be on a stable antidepressant therapeutic regimen, or not receiving treatment for 4 weeks prior to study enrollment and agree to continue this regimen throughout the study period.
8. In good general health, as evidenced by medical history.
9. For persons of child-bearing potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
10. Agreement to adhere to Lifestyle Considerations (i.e. must continue with any existing treatments) throughout study duration.
11. For persons of child-bearing potential: must take a pregnancy test at the screening visit, with results confirmed as negative by study staff.

Exclusion Criteria:

An individual will be excluded from participation in this study if they meet any of the following criteria, as determined from a review of medical records prior to screening or at the screening visit:

1. Pregnancy;
2. History of psychotic or bipolar disorder or depression with psychotic features;
3. Significant borderline personality disorder;
4. Significant comorbid obsessive-compulsive or post-traumatic stress disorder;
5. Previously diagnosed Intellectual Disability or Autism Spectrum Disorder;
6. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal;
7. Clinically significant suicidality;
8. Any history of tDCS;
9. Any history of ECT;
10. History of TMS (greater than 15 sessions) without a clinically meaningful response.
11. History of ketamine (greater than 4 sessions) without a clinically meaningful response;
12. Chronic depression (defined as of over 5 years duration);
13. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma with persistent symptoms;
14. Untreated or insufficiently treated endocrine disorder;
15. Contraindication to receiving tDCS (e.g., ferromagnetic implant, history of seizure, known brain lesion);
16. Treatment with an investigational drug or other intervention within the study period;
17. Unstable symptoms between screening and baseline as defined by a ≥ 30% change in MADRS score;
18. Require a benzodiazepine with a dose > lorazepam 2 mg/day
19. Has started a new psychotherapeutic process in the past 3 months from screening;
20. Use of potentially irritant topical treatments (ex: retinoids, alpha hydroxy acids)
21. Aesthetic procedure the area of the forehead directly below the stimulation area within the last 6 months (laser, fillers, surgery, etc.)
22. Any active dermatological condition on face or scalp that would in the opinion of the PI represent a contraindication to the treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility (Recruitment) | From baseline clinical assessment prior to treatment, to 6 weeks after first treatment.
  Recruitment rate will be measured as the number of patients enrolled by the conclusion of the study, reported as a whole number.
Feasibility (Retention) | From baseline clinical assessment prior to treatment, to 6 weeks after first treatment.
  Retention rate will be measured as the percentage of enrolled patients who complete all study visits, reported as a percentage.
Feasibility (Adherence) | From baseline clinical assessment prior to treatment, to 6 weeks after first treatment.
  The proportion of completed sessions relative to the total prescribed sessions, expressed as a percentage.
Safety | From baseline clinical assessment prior to treatment, to 6 weeks after first treatment.
  Safety will be measured by the number of serious adverse events (SAEs).
Tolerability | From baseline clinical assessment prior to treatment, to 6 weeks after first treatment.
  Tolerability will be measured by the number of adverse events (AEs).

SECONDARY OUTCOMES:
Biomarker Discovery: Short-Interval Intracortical Inhibition (SICI) via TMS-EMG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 6 weeks after first treatment.
  TMS-EMG will be used to evaluate changes in SICI.
  Unit of Measurement: Amplitude or percentage inhibition.
Biomarker Discovery: Intracortical Facilitation (ICF) via TMS-EMG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 6 weeks after first treatment.
  TMS-EMG will be used to evaluate changes in intracortical facilitation
  Unit of Measurement: Amplitude or percentage facilitation.
Biomarker Discovery: Cortical Silent Period (CSP) via Transcranial Magnetic Stimulation-Electromyography (TMS-EMG) | From baseline neurophysiological assessment prior to treatment, to during treatment, to 6 weeks after first treatment.
  TMS-EMG will be used to assess changes in the cortical silent period (CSP).
  Unit of Measurement: Duration (milliseconds).
Biomarker Discovery: TMS-Evoked Potential (TEP) Component Amplitudes via TMS-EEG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 6 weeks after first treatment.
  TMS-EEG will be used to evaluate changes in TMS-evoked potential (TEP) component amplitudes.
  Unit of Measurement: Voltage (µV).
Biomarker Discovery: Significant Current Density (SCD) via TMS-EEG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 6 weeks after first treatment.
  TMS-EEG will be used to evaluate changes in significant current density (SCD).
  Unit of Measurement: Current density (A/m²).
Biomarker Discovery: Biomarker Discovery: Significant Current Scattering (SCS) via TMS-EEG | From baseline neurophysiological assessment prior to treatment, to during treatment, to 6 weeks after first treatment.
  TMS-EEG will be used to evaluate changes in significant current scattering (SCS).
  Unit of Measurement: Scattering coefficient (unitless).
Biomarker Discovery: Resting-State Electroencephalography (rsEEG) | From baseline neurophysiological assessment prior to treatment, to during treatment, to 6 weeks after first treatment.
  rsEEG will be used to analyze changes in brain activity patterns at rest.
  Unit of Measurement: Frequency (Hz) and amplitude (µV).
Changes from pre-treatment depressive symptomatology in post-treatment | From baseline clinical assessment prior to treatment, to 6 weeks after first treatment.
  Changes in depressive symptoms will be assessed using the Montgomery-Åsberg Depression Rating Scale (MADRS), which ranges from 0 to 60, with higher scores indicating more severe depression. A decrease in the MADRS score will be interpreted as an improvement in symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Interventional Psychiatry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No